CLINICAL TRIAL: NCT05256745
Title: RAGE Inhibition to Decrease Cancer Therapy Related Cardio Toxicity in Women With Early Breast Cancer
Brief Title: RAGE Inhibition to Decrease Cardiotoxicity in Women With Early Breast Cancer
Acronym: RAGE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003782
Record Dates: First submitted 2022-01-03; First posted 2022-02-25 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Cancer Related Cognitive Decline; Non-metastatic Breast Cancer
MeSH Terms: interventions — azeliragon; Cyclophosphamide; Docetaxel; Carboplatin; Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: TTP488 (Azeliragon) co-administered with dose dense paclitaxel (ddAC/ddT) (Experimental): Cohort 1: On day 7 of cycle 3, twelve capsules of azeliragon taken daily for 6 days, and then four capsules of Azeliragon each day continuously through the end of that cycle of chemotherapy, extending into Cycle 4 Day 2 (C4D2).
  Interventions: Drug: TTP488; Drug: ddAC/ddT
- Cohort 2: TTP488 (Azeliragon) co-administered with TC (Experimental): TC: docetaxel and cyclophosphamide
  Cohort 2a (6 cycles): Cycle 5 Day 14 (C5D14), take twelve capsules of azeliragon daily for 6 days, then four capsules of Azeliragon each day continuously through the end of that cycle of chemotherapy, extending into Cycle 6 Day 2 (C6D2).
  Cohort 2b (4 cycles): Cycle 3 Day 14 (C3D14), take twelve capsules of azeliragon daily for 6 days, then four capsules of Azeliragon each day continuously through the end of that cycle of chemotherapy, extending into Cycle 4 Day 2 (C4D2).
  Interventions: Drug: TTP488; Drug: TC
- Cohort 3: TTP488 (Azeliragon) co-administered with TCHP (Experimental): TCHP: docetaxel, carboplatin, trastuzumab, and pertuzumab Cohort 3: Cycle 5 Day 14 (C5D14), take twelve capsules of azeliragon daily for 6 days, then four capsules of Azeliragon each day continuously through the end of that cycle of chemotherapy, extending into Cycle 6 Day 2 (C6D2).
  Interventions: Drug: TTP488; Drug: TCHP
- Cohort 4: TTP488 (Azeliragon) co-administered with chemotherapy regimen that includes ddAC (Experimental): given at the end of the chemotherapy plan [can include: (1)weekly carboplatin + paclitaxel + pembrolizumab followed by pembrolizumab + dose dense doxorubicin and cyclophosphamide; (2) weekly carboplatin + paclitaxel followed by dose dense doxorubicin and cyclophosphamide; (3) weekly or dose dense paclitaxel followed by dose dense doxorubicin and cyclophosphamide]
  Cohort 4: On day 7 of cycle 3, twelve capsules of azeliragon taken daily for 6 days, and then four capsules of Azeliragon each day continuously through the end of that cycle of chemotherapy, extending into Cycle 4 Day 2 (C4D2).
  Interventions: Drug: TTP488; Drug: Chemotherapy regimen that includes ddAC

INTERVENTIONS:
Drug: TTP488 — Each Azeliragon capsule is 5mg, and is to be taken in the morning with food as indicated in each cohort.
  Other Names: Azeliragon
Drug: ddAC/ddT — Dose dense doxorubicin plus cyclophosphamide followed by paclitaxel (ddAC/ddT) for 8 cycles, administered per USPI (Unites States Prescribing Information) Label
  Other Names: Dose dense doxorubicin plus cyclophosphamide, dose dense paclitaxel
  Arms: Cohort 1: TTP488 (Azeliragon) co-administered with dose dense paclitaxel (ddAC/ddT)
Drug: TC — Docetaxel plus cyclophosphamide (TC) for 4-6 cycles, administered per USPI (Unites States Prescribing Information) Label
  Other Names: Docetaxel plus cyclophosphamide
  Arms: Cohort 2: TTP488 (Azeliragon) co-administered with TC
Drug: TCHP — Docetaxel, carboplatin, trastuzumab, and pertuzumab (TCHP)for 6 cycles, administered per USPI (Unites States Prescribing Information) Label
  Other Names: Docetaxel, carboplatin, trastuzumab, and pertuzumab
  Arms: Cohort 3: TTP488 (Azeliragon) co-administered with TCHP
Drug: Chemotherapy regimen that includes ddAC — can include: (1) weekly carboplatin + paclitaxel + pembrolizumab followed by pembrolizumab + dose dense doxorubicin and cyclophosphamide; (2) weekly carboplatin + paclitaxel followed by dose dense doxorubicin and cyclophosphamide; (3) weekly or dose dense paclitaxel followed by dose dense doxorubicin and cyclophosphamide, administered per USPI (Unites States Prescribing Information) Label
  Other Names: Dose dense doxorubicin plus cyclophosphamide
  Arms: Cohort 4: TTP488 (Azeliragon) co-administered with chemotherapy regimen that includes ddAC

SUMMARY:
This is a pilot study to evaluate the effects of azeliragon to decrease cardiac toxicity from chemotherapy and the safety of azelirgaon when given with chemotherapy. The Investigators hypothesize that there will be no significant interaction with Azeliragon and chemotherapy and that targeting the RAGE pathway will decrease anthracycline related cardiotoxicity and chemotherapy related cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have clinical or pathologic stage I-III, histologically confirmed breast cancer, with any ER (estrogen-receptor), PR (progesterone receptors), or HER2 (human epidermal growth factor receptor 2) status who are planned to receive chemotherapy in the adjuvant or neoadjuvant setting.

   a. Chemotherapy regimens administered per USPI (United States Prescribing Information) label: i. Dose dense doxorubicin plus cyclophosphamide followed by paclitaxel (ddAC/ddT) for 8 cycles ii. Docetaxel plus cyclophosphamide (TC) for 4-6 cycles iii. Docetaxel, carboplatin, trastuzumab, and pertuzumab (TCHP)for 6 cycles iv. Chemotherapy regimen that includes ddAC, given at the end of the chemotherapy plan [can include: (1)weekly carboplatin + paclitaxel + pembrolizumab followed by pembrolizumab + dose dense doxorubicin and cyclophosphamide; (2) weekly carboplatin + paclitaxel followed by dose dense doxorubicin and cyclophosphamide; (3) weekly or dd paclitaxel followed by dose dense doxorubicin and cyclophosphamide]
2. Patients must have had no prior chemotherapy/radiotherapy/or systemic therapy for early stage breast cancer, or any other malignancy
3. Age ≥18 years.
4. ECOG (Eastern Cooperative Oncology Group) performance status ≤2 (Karnofsky ≥60%, see Appendix D).
5. Patients must have normal organ and marrow function as defined below:

   1. Leukocytes ≥3,000/mcL (microliter)
   2. Absolute neutrophil count ≥1,500/mcL
   3. Platelets ≥100,000/mcL
   4. Total bilirubin ≤ 2.0 x institutional upper limit of normal (ULN)
   5. AST(SGOT) (aspartate transaminase)/ALT(SGPT) (alanine aminotransferase) ≤1.5 × institutional ULN
   6. Glomerular filtration rate (GFR) ≥60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
6. Human immunodeficiency virus (HIV)-infected patients on effective antiretroviral therapy with undetectable viral load within 6 months are eligible for this trial. If evidence of chronic hepatitis B virus (HBV) infection, HBV viral load must be undetectable on suppressive therapy if indicated. If history of hepatitis C virus (HCV) infection, must be treated with undetectable HCV viral load.
7. No pre-existing neurodegenerative disease or impairment, including history of CVA (cerebrovascular accident), or head injury.
8. No psychiatric disorders which could interfere with their ability to consent. (Allowed psychiatric disorders may include but are not limited to: anxiety, depression, obsessive compulsive disorder, ADHD; as long as the disorder does not affect the ability to consent). Any other psychiatric disorders should be discussed with the Principal Investigator (PI) and will be allowed at the discretion of the PI.
9. The effects of azeliragon on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
10. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who have had prior chemotherapy, radiotherapy, systemic therapy, or hormonal therapy
2. Patients with Stage IV breast cancer
3. Patients who are receiving any other investigational agents.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to azeliragon, or the standard of care chemotherapy assigned, including: docetaxel, cyclophosphamide, carboplatin, doxorubicin, paclitaxel, trastuzumab, pertuzumab, pembrolizumab.
5. Patients receiving any medications or substances that are strong CYP2C8 inhibitors are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product. Subjects who discontinue a strong CYP2C8 inhibitor must have discontinued the drug for at least 5 days or 5 half-lives of the drug, whichever is longer, before the first dose of study drug.
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, neurogenerative disease/impairment, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Pregnant women are excluded from this study as the risks of azeliragon to a fetus are unknown. There is unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with azeliragon; breastfeeding should be discontinued if the mother is treated with azeliragon. These potential risks may also apply to other agents used in this study.
8. History of cancer within the last 5 years except adequately treated cervical carcinoma-in-situ, or cutaneous basal cell or squamous cell cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of unacceptable toxicity | 1 cycle (Cohort 1 and 4 each cycle is 14 days; Cohort 2 and 3 each cycle is 21 days)
  Any Adverse Event (AE) considered unrelated to chemotherapy, underlying disease, disease progression, intercurrent illness or concomitant medications/therapies resulting in the inability to tolerate the cycle of chemotherapy
Incidence of severe AE graded according to the CTCAE v.5 | 1 cycle (Cohort 1 and 4 each cycle is 14 days; Cohort 2 and 3 each cycle is 21 days)
Incidence of chemotherapy dose interruption, dose modification, dose discontinuation | 1 cycle (Cohort 1 and 4 each cycle is 14 days; Cohort 2 and 3 each cycle is 21 days)
Change in Troponin level | Cohort 1 and 4: cycle 3 and cycle 4, day 1 and day 2 of 14 day cycle; Cohort 2 and 3:cycle 5 and cycle 6, day 1 and day 2 of 21 day cycle]
  • Change in troponin levels after administration of chemotherapy, in those treated with and without azeliragon.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) assessment: Cmax | Cohort 1 and 4: cycle 3 and cycle 4, day 1 and day 2 of 14 day cycle; Cohort 2 and 3:cycle 5 and cycle 6, day 1 and day 2 of 21 day cycle
  Maximum observed serum concentration
Pharmacokinetic (PK) assessment: tmax | Cohort 1 and 4: cycle 3 and cycle 4, day 1 and day 2 of 14 day cycle; Cohort 2 and 3:cycle 5 and cycle 6, day 1 and day 2 of 21 day cycle
  Time of maximum observed serum concentration
Pharmacokinetic (PK) assessment: AUC0-last | Cohort 1 and 4: cycle 3 and cycle 4, day 1 and day 2 of 14 day cycle; Cohort 2 and 3:cycle 5 and cycle 6, day 1 and day 2 of 21 day cycle
  Area under the serum concentration-time curve from time zero to the last quantifiable timepoint
Pharmacokinetic (PK) assessment: AUC0-INF | Cohort 1 and 4: cycle 3 and cycle 4, day 1 and day 2 of 14 day cycle; Cohort 2 and 3:cycle 5 and cycle 6, day 1 and day 2 of 21 day cycle
  Area under the serum concentration-time curve from time zero extrapolated to infinity
Pharmacokinetic (PK) assessment: AUC0-tau | Cohort 1 and 4: cycle 3 and cycle 4, day 1 and day 2 of 14 day cycle; Cohort 2 and 3:cycle 5 and cycle 6, day 1 and day 2 of 21 day cycle
  Area under the serum concentration-time curve from time zero to the end of the dosing interval
Pharmacokinetic (PK) assessment: t1/2 | Cohort 1 and 4: cycle 3 and cycle 4, day 1 and day 2 of 14 day cycle; Cohort 2 and 3:cycle 5 and cycle 6, day 1 and day 2 of 21 day cycle]
  Terminal elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: Candace Mainor, MD, Principal Investigator — Georgetown University
Locations (3):
- United States (3):
  - Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: No